CLINICAL TRIAL: NCT05722886
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations
Brief Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial) - Master Screening Protocol
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Manchester (Other); University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Hoffmann-La Roche (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004; IRAS ID: 1004057 (Other: IRAS)
Record Dates: First submitted 2022-11-24; First posted 2023-02-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Haematological Malignancy; Solid Tumour
Keywords: Adult; Alectinib; ALK Tyrosine Kinase Receptor; Antineoplastic Agents; Atezolizumab; BRAF Kinase; Cancer; Child; CMMRD; Cobimetinib; Entrectinib; Genes, HER2; Immune Checkpoint Inhibitors; Immunological; Lymphoproliferative Disorders; Malignancy; Malignant Neoplasms; MSI; Molecular Targeted Therapy; Mutation; Neoplasms by Histologic Type; Neoplasms by Site; Paediatric; Pertuzumab; Precision Medicine; Protein Kinase Inhibitors; Rare; ROS1 protein, human; TMB; Trastuzumab; Tumour-agnostic; Vemurafenib; Young adult; Capmatinib; MET
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms by Site | interventions — alectinib; atezolizumab; entrectinib; Trastuzumab; pertuzumab; Vemurafenib; cobimetinib; capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Arm 1: Alectinib (Experimental): This alectinib treatment arm is for adult, paediatric and TYA patients with ALK-positive cancers.
  Interventions: Drug: Alectinib
- Treatment Arm 2: Atezolizumab (Experimental): This atezolizumab treatment arm is for adult, paediatric and TYA patients with cancers with high tumour mutational burden (TMB) or microsatellite instability high (MSI-high) or proven (previously diagnosed) constitutional mismatch repair deficiency (CMMRD).
  Interventions: Drug: Atezolizumab
- Treatment Arm 3: Entrectinib (Experimental): This entrectinib treatment arm is for adult, paediatric and TYA patients with ROS1 gene fusion-positive cancers.
  Interventions: Drug: Entrectinib
- Treatment Arm 4: Trastuzumab in combination with pertuzumab (Experimental): This trastuzumab and pertuzumab treatment arm is for adult, paediatric and TYA patients with cancers with HER2 amplification or activating mutations.
  Interventions: Drug: Trastuzumab in combination with pertuzumab
- Treatment Arm 5: Vemurafenib in combination with cobimetinib (Experimental): This vemurafenib and cobimetinib treatment arm is for BRAF V600 mutation-positive cancers occurring in adults only.
  Interventions: Drug: Vemurafenib in combination with cobimetinib
- Treatment Arm 6: Capmatinib (Experimental): This capmatinib treatment arm is for adult patients with cancers harbouring MET dysregulations.
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Alectinib — Adult patients will be administered alectinib orally at a dose of 600 mg (four 150 mg capsules) twice daily.
  Paediatric patients with a body weight ≥40 kg and who are able to swallow the capsules will be administered alectinib orally at a dose of 600 mg (four 150 mg capsules) twice daily.
  Each cycle of treatment will consist of 28 days and patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Alecensa
  Arms: Treatment Arm 1: Alectinib
Drug: Atezolizumab — Adult patients will receive 1200 mg of atezolizumab intravenously every 21 days.
  Paediatric patients will receive atezolizumab at a dose of 15 mg/kg (maximum 1200 mg) every 21 days.
  Patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Tecentriq
  Arms: Treatment Arm 2: Atezolizumab
Drug: Entrectinib — Adult and paediatric patients with body surface area (BSA) ≥1.51 m^2 will receive entrectinib orally at a dose of 600 mg daily dose (three 200 mg capsules per day).
  Paediatric patients with BSA <1.51 m^2 will receive a dose adjusted for BSA. Each cycle of treatment will consist of 28 days and patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Rozlytrek
  Arms: Treatment Arm 3: Entrectinib
Drug: Trastuzumab in combination with pertuzumab — The initial loading dose of trastuzumab is 8 mg/kg body weight followed thereafter by a maintenance dose of 6 mg/kg body weight administered intravenously every 21 days.
  The initial loading dose of pertuzumab is 840 mg followed thereafter by a maintenance dose of 420 mg administered intravenously every 21 days. Paediatric patients will receive a dose of pertuzumab adjusted by body weight.
  Patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Herceptin in combination with Perjeta
  Arms: Treatment Arm 4: Trastuzumab in combination with pertuzumab
Drug: Vemurafenib in combination with cobimetinib — Patients will receive vemurafenib at a dose of 960 mg (four tablets of 240 mg) orally on a twice daily schedule throughout a 28-day cycle.
  Patients will receive cobimetinib at a dose of 60 mg (three tablets of 20 mg) to be taken orally, once daily for 21 consecutive days (days 1 to 21 in each 28-day cycle); followed by a 7-day break.
  Patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Zelboraf in combination with Cotellic
  Arms: Treatment Arm 5: Vemurafenib in combination with cobimetinib
Drug: Capmatinib — Patients will be administered capmatinib orally at a daily dose of 800 mg consisting of 400 mg (two 200 mg tablets) twice daily. Each cycle of treatment will consist of 28 days and patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Tabrecta
  Arms: Treatment Arm 6: Capmatinib

SUMMARY:
DETERMINE is an open-label phase II/III trial. It will look at targeted treatments in rare cancers or common cancers with rare genetic change (mutation). Patients must have a cancer with an identified mutation. This could be found during routine testing or as part of another research programme. The DETERMINE trial will recruit adults, teenagers and children. If a drug is found to benefit a new patient group, the study team will work with the NHS and the Cancer Drugs Funds to see if these drugs can be available for patients in the future. This clinicaltrials.gov record refers to the Overall Trial Protocol (Master Screening Record), additional records will be added to clinicaltrials.gov for each treatment arm.

DETAILED DESCRIPTION:
DETERMINE is an umbrella-basket platform trial to evaluate the efficacy of licensed targeted therapies in rare* adult, paediatric and teenage/young adult (TYA) cancers with actionable genomic alterations, including common cancers with rare actionable alterations.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients (includes paediatric and TYA cancers) or common cancers with rare alterations.

The number of treatment arms opened will depend on the number of licensed medicines identified for inclusion. Each trial cohort has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

This clinicaltrials.gov record refers to the Overall Trial Protocol (Master Screening Record), please refer to the references section for links to the individual treatment arm records.

The main aims of the clinical trial arms are:

* To describe the anti-cancer activity of licensed targeted drugs outside their licensed indication.
* To assess the safety and adverse event (AE) profile of licensed, targeted anti-cancer drugs in the target population.
* To understand biological mechanisms for response and resistance to targeted therapies.
* To evaluate the quality of life (QoL) of target populations receiving the licensed, targeted anti-cancer drugs.

This Master Screening Record will capture the number of patients with a cancer containing the appropriate genetic alteration that have been successfully allocated and consented to each arm. The trial results (according to the protocol defined outcome measures) will be reported per-arm for each treatment arm.

The ultimate aim is to translate positive clinical findings to the NHS to provide new treatment options for rare adult, paediatric and TYA cancers.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA OUTLINED BELOW AND WITHIN THE SPECIFIC TREATMENT ARM APPENDIX TO WHICH THEY ARE ENROLLED.

Core Inclusion Criteria:

1. Any patient (adult patients or children and TYA as defined in each treatment arm appendix) with histologically proven locally advanced or metastatic cancer (solid tumour or haematological malignancy) who has:

   1. exhausted (or declined) standard-of-care treatment options.
   2. or for whom no effective standard treatment is available.
   3. and whose disease has progressed or is refractory. Exceptional circumstances may apply as described in the protocol.
2. Diagnosis of a rare cancer harbouring an actionable genomic alteration, or common cancer types with rare actionable genomic alterations, that has been identified using a validated next-generation sequencing method and for which there is a relevant open treatment arm within the DETERMINE trial.
3. Life expectancy of at least three months.
4. Patients are able to provide written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up. For patients under 16 years old, the parent or legal guardian will be asked to provide written informed consent and the patient will be asked to provide age-appropriate assent (written or verbal, commensurate with age and level of understanding).
5. Patients with objectively evaluable or measurable disease, according to an assessment method appropriate for their cancer type.
6. Patients must provide a fresh tissue biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow and/or trephine or lymph node biopsy samples may be taken.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (ECOG performance status 2 may be considered on an individual basis) (adults), Karnofsky score ≥50% (TYA) or Lansky Play scales ≥50% (<12 years). Please see specific treatment arm appendices for any variations on this criterion and for definitions of adult and paediatric populations. Note: Paediatric patients: patients with Central Nervous System (CNS) tumours and a stable neurological deficit may be eligible with a performance status below 50%, at the discretion of the Investigator. In such cases, the deficit must be stable for at least 7 days prior to trial enrolment and be assessed by the local investigator as due to tumour or due to a post-surgical AE.
8. Women of childbearing potential are eligible provided that they meet the following criteria:

   * Have a negative serum or urine pregnancy test before enrolment and
   * Agree to the birth control methods and duration of use of those methods, as specified in each treatment arm appendix.
9. Male patients with partners of childbearing potential are eligible provided that they agree to the birth control methods and duration of use of those methods, as specified in each treatment arm appendix.

Core exclusion criteria:

1. Ongoing AEs Common Terminology Criteria of Adverse Events (CTCAE) Grade ≥2 attributable to previous anti-cancer treatments. Exceptions to this are any clinically stable AEs, which in the opinion of the Investigator should not exclude the patient.
2. At high medical risk, in the opinion of the Investigator, because of non-malignant systemic disease (including active uncontrolled infection).
3. Female patients who are pregnant, breastfeeding or planning to become pregnant or male patients with a partner who is a woman of childbearing potential and is planning to become pregnant during the trial or following the last dose of IMP, as specified in each treatment arm appendix.
4. Is (or plans to be) a patient in another interventional clinical trial, whilst taking part in this trial. Participation in an observational trial which does not involve administration of an Investigational Medicinal Product (IMP) and which, in the opinion of the local Investigator, would not place an unacceptable burden on the patient would be acceptable e.g. sample collection* or QoL studies.

   *for paediatric patients participating in other studies involving tissue/circulating tumour (ct) DNA/other blood collection, consideration would need to be given to the total blood volumes collected (as per the European Medicines Agency blood volume limits for children).
5. Co-administration of anti-cancer therapies other than those administered in this trial (with the exception of lifelong hormone suppression such as luteinising hormone agonists/analogues in prostate cancer).
6. Radiotherapy (except for palliative reasons) or chemotherapy, endocrine therapy (except when given for conditions other than malignant disease; e.g. thyroid replacement for hypothyroidism, hydrocortisone for cortisol deficiency/panhypopituitarism), nitrosoureas, mitomycin-C, immunotherapy and molecularly targeted agents or other IMPs within 4 weeks or 5 half-lives (whichever is the shorter).
7. Rapidly progressing or symptomatically deteriorating brain metastases. Patients with previously treated brain metastases are eligible, provided the patient has not experienced a seizure or had a clinically significant change in neurological status within the 14 days (for adult patients) or 7 days (for paediatric patients) prior to the start of IMP administration. Such patients must be non-dependent on steroids or on a stable or reducing dose of steroid treatment for at least 14 days (or 7 days for paediatric patients) prior to the start of IMP administration. Primary brain or CNS malignancies are allowed providing the patient is clinically stable (if requiring corticosteroids must be at stable or decreasing doses for at least 14 days for adults and 7 days for paediatric patients prior to the start of IMP administration). Patients who have received brain irradiation must have completed whole-brain radiotherapy and/or stereotactic radiosurgery at least 14 days prior to the start of IMP administration.
8. Any other condition which, in the opinion of the local Investigator, would not be in the best interests of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who consent to each arm. | Up to 5 years.
  This is a master screening entry with sub-study entries to capture the results of each arm. As such a primary outcome measure for this entry is not relevant, however this entry will be used to report the number of patients with a cancer containing the appropriate genetic alteration that have been successfully allocated and consented to each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (27):
- United Kingdom (27):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cardiff Children's Hospital, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Royal Hospital for Children Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Hospital, Liverpool
  - University College London Hospital, London
  - Guy's Hospital, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Great North Children's Hospital, Newcastle
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Sheffield's Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests made within 5 years from last patient last visit for each of the treatment arms will be considered (refer to individual treatment arm records); requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk

REFERENCES:
- See also: Overview of the DETERMINE trial. — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 01 (alectinib) (NCT05770037) — https://clinicaltrials.gov/ct2/show/NCT05770037
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 02 (atezolizumab) (NCT05770102) — https://clinicaltrials.gov/ct2/show/NCT05770102
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 03 (entrectinib) (NCT05770544) — https://clinicaltrials.gov/ct2/show/NCT05770544
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 04 (trastuzumab in combination with pertuzumab) (NCT05786716) — https://clinicaltrials.gov/ct2/show/NCT05786716
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 05 (vemurafenib in combination with cobimetinib) (NCT05768178) — https://clinicaltrials.gov/ct2/show/NCT05768178
- See also: ClinicalTrials.gov record for DETERMINE Trial Treatment Arm 06 (capmatinib) (NCT06988475) — https://clinicaltrials.gov/study/NCT06988475